CLINICAL TRIAL: NCT06288035
Title: Oral Dexamethasone at Night to Prevent Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy: A Protocol for Randomized Clinical Trial
Brief Title: Oral Dexamethasone for Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R.21.02.1191
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a parallel, two-arm, randomized (1:1), controlled, single-center non-inferiority trial. Adults (≥18 years) with ASA physical status I-III scheduled for elective laparoscopic cholecystectomy will be eligible for inclusion. The participants will be randomized to receive either 8 mg of IV Dexamethasone at the time of induction of anesthesia or 8 mg of oral Dexamethasone at night before surgery. The primary outcome will be the incidence of postoperative nausea and vomiting. 814 patients are intended to be recruited for this non-inferiority trial.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-night oral dexamethasone (Experimental): Patients in the intervention group will receive oral 8 mg dexamethasone at night before surgery. The time of dexamethasone administration will be recorded.
  Interventions: Drug: Dexamethasone Oral
- At-induction dexamethasone (Active Comparator): Patients in the control group will receive intravenous 8 mg dexamethasone just before or at the induction of anesthesia. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensations in injection.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone Oral — Patients in the intervention group will receive oral 8 mg dexamethasone at night before surgery. The time of dexamethasone administration will be recorded.
  Arms: At-night oral dexamethasone
Drug: Dexamethasone — Patients in the control group will receive intravenous 8 mg dexamethasone just before or at the induction of anesthesia. The dexamethasone ampule will be diluted in a 10 ml syringe and given in at least one minute to avoid unpleasant sensations in injection.
  Arms: At-induction dexamethasone

SUMMARY:
Postoperative nausea and vomiting (PONV) are common complications after laparoscopic cholecystectomy. This study aims to evaluate the efficacy of the administration of prophylactic oral dexamethasone at night before surgery in preventing PONV after elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Background:

Postoperative nausea and vomiting (PONV) are common complications after laparoscopic cholecystectomy. This study aims to evaluate the efficacy of the administration of prophylactic oral dexamethasone 12 hours before induction of anesthesia in preventing PONV after elective laparoscopic cholecystectomy, as it reaches its peak effect at 2-12 hours and lasts for 72 hours after oral administration.

Methods:

This is a parallel, two-arm, randomized (1:1), controlled, single-center non-inferiority trial. Adults (≥18 years) with ASA physical status I-III scheduled for elective laparoscopic cholecystectomy will be eligible for inclusion. The participants will be randomized to receive either 8 mg of IV Dexamethasone at the time of induction of anesthesia or 8 mg of oral Dexamethasone 12 hours before induction of anesthesia. The primary outcome will be the incidence of postoperative nausea and vomiting. A total of 814 patients are intended to be recruited for this non-inferiority trial.

Discussion:

The current randomized trial is exploring the non-inferiority and feasibility of oral dexamethasone at night to reduce the PONV after laparoscopic cholecystectomy when compared to the standard of care - intravenous dexamethasone at the time of induction. Additionally, the investigators suppose oral dexamethasone at night is easier to administer, avoids polypharmacy at the time of induction of anesthesia, avoids the unpleasant sensation of intravenous injection, and is at a lower cost for a one-day surgery.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive adults (older than 18 years) with ASA physical status I-III undergoing elective laparoscopic cholecystectomy surgery.

Exclusion Criteria:

* steroids or antiemetics within 1 week of surgery
* chronic opioid therapy
* history of allergy to any of the study drug
* serum creatinine > 1.4 mg/dl
* liver enzymes > triple the normal limits
* pregnancy
* patient refusal
* and psychiatric or neurologic diseases or socioeconomic status that would hinder the postoperative quality of recovery questionnaire
* laparoscopic surgery is converted to open surgery after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea or vomiting (PONV) | 24 hours after surgery
  incidecne of PONV

SECONDARY OUTCOMES:
Rescue antiemetic | 24 hours after surgery
  need for rescue antiemetic for 24 hours after surgery (Dichotomous yes/no outcome)
Early PONV | within 6 hours after surgery
  (Dichotomous yes/no outcome)
Late PONV | 6 - 24 hours after surgery
  (Dichotomous yes/no outcome)
Visual Analogue Scale (VAS) at the time of discharge from PACU | within 2 hours at the time of discharge from PACU
  On VAS scale as numerical outcome
VAS at the time of discharge from hospital | after 24 hours at the time of discharge from the hospital
  On VAS scale as numerical outcome
Postoperative fatigue | after 24 hours at the time of discharge from the hospital
  on a 10-point scale
Postoperative quality of recovery | after 24 hours at the time of discharge from the hospital
  using the QoR-15 questionnaire
Post-Discharge Nausea and Vomiting (PDNV) | 72 hours after surgery.
  evaluated by telephone as a binary outcome

OTHER OUTCOMES:
Surgical Site Infection (at follow-up) | within 2 weeks - on the follow-up
  as evaluated by the surgeon
Itching or burning sensation on dexamethasone injections | during injection of the dexamethoasone
  Dichotomous yes/no outcome

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Faculty of Medicine, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available with the principal investigator on a reasonable request after approval of the local IRB.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year after the completion of the study
Access Criteria: Will be reported after completion of the study.